CLINICAL TRIAL: NCT05725122
Title: Stone Clearance in Patients With Upper Ureteric Stones Using Extracorporeal Shock Wave Lithotripsy Compared With Extracorporeal Shock Wave Lithotripsy Combined With Tamsulosin Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, Principal Investigator, Services Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S23
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis | interventions — Lithotripsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWL alone (Active Comparator): Extracorporeal shock wave lithotripsy will be given to the patient
  Interventions: Procedure: Extracorporeal shock wave lithotripsy
- ESWL combined with tamsulosin therapy (Active Comparator): Extracorporeal shock wave lithotripsy combined with tamsulosin therapy will be given to the patient
  Interventions: Procedure: Extracorporeal Shock Wave Lithotripsy combined with Tamsulosin Therapy.

INTERVENTIONS:
Procedure: Extracorporeal shock wave lithotripsy — Extracorporeal shock wave lithotripsy will given to the patients
  Arms: ESWL alone
Procedure: Extracorporeal Shock Wave Lithotripsy combined with Tamsulosin Therapy. — Extracorporeal Shock Wave Lithotripsy combined with Tamsulosin Therapy will be given to the patients
  Arms: ESWL combined with tamsulosin therapy

SUMMARY:
Extracorporeal shock wave lithotripsy (ESWL) is the least invasive and effective treatment for upper ureteric stones with a stone clearance rate of 60-90%. Tamsulosin is an alpha-blocker widely used in urological practice to relax smooth muscle of the prostate and bladder neck. Its role as part of medical expulsion therapy for the treatment of patients with kidney and ureteric stones has proved to be of considerable success. However, its role in clearing upper ureteric stones as an adjunct to ESWL is controversial. Therefore, this study will be conducted to evaluate its role in stone clearance along with extracorporeal shock wave lithotripsy in patients with upper ureteric stones

ELIGIBILITY:
Inclusion Criteria:

* single upper ureteric stone
* size ranging from 6-15 mm
* stones history less than 6 months

Exclusion Criteria:

* Patients with urinary tract infection
* multiple ureteric stones,
* presence of a ureteric stricture distal to the stone,
* previous unsuccessful ESWL,
* concomitant use of calcium channel blockers or alpha-adrenergic antagonists
* patients with abnormal coagulation profile

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
stone clearance | 4 weeks
  Number of patients cleared from ureteric stones

CONTACTS AND LOCATIONS:
Locations (1):
- services Institute of Medical Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided